CLINICAL TRIAL: NCT02858713
Title: Can an App Supporting Psoriasis Patients Improve Adherence to Topical Treatment? A Single-blind Randomized Controlled Trial
Brief Title: Adherence in Topical Treatment of Psoriasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Mathias Tiedemann Svendsen, MD, PhD, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2016-002143-42
Record Dates: First submitted 2016-08-03; First posted 2016-08-08 (Estimated); Results first posted 2019-06-03 (Actual); Last update posted 2019-06-03 (Actual); Status verified 2019-02

CONDITIONS: Adherence
Keywords: psoriasis
MeSH Terms: conditions — Psoriasis | interventions — betamethasone dipropionate, calcipotriol drug combination

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- App as intervention + Enstilar© (Experimental): Patients prescribed Calcipotriene + Betamethasone Dipropionatecutaneous foam receive the intervention EM with app for smartphone and conventional instruction from a nurse in the consultation.
  Interventions: Drug: Calcipotriene + Betamethasone Dipropionate; Device: App
- Conventional instructions + Enstilar© (No Intervention): Patients receive conventional instructions from a nurse in the consultation in how to use prescribed Enstilar© with EM.

INTERVENTIONS:
Drug: Calcipotriene + Betamethasone Dipropionate — Participants received Calcipotriene + Betamethasone Dipropionate once daily when needed for the entire study period.
  Other Names: Enstilar
  Arms: App as intervention + Enstilar©
Device: App — App named MyPso SmarTopTM Version 1.0 (LEO Pharma) was used for 28 days by participants in the intervention arm.
  Other Names: Mypso app
  Arms: App as intervention + Enstilar©

SUMMARY:
Medical adherence to topical corticosteroid products in psoriasis patients is a main determinant for poor treatment effect.

The investigators aim to test if a multifaceted intervention delivered in an app (MyPso QualityCareTM owned by Leo Pharma) for smartphones combined with an Electronic Monitor (EM) (Teslo) can improve medical adherence among psoriasis patients treated with a topical calcipotriol/betamethasone dipropionate foam combination (Cal/BD) (Enstilar©).

The study is classified as a phase 4 study, since it is studied if improved use of Enstilar© results in improved treatment outcomes.

Link to published study protocol:

https://bmcdermatol.biomedcentral.com/articles/10.1186/s12895-018-0071-3

Link to published results from the study:

https://onlinelibrary.wiley.com/doi/abs/10.1111/bjd.16667

DETAILED DESCRIPTION:
Material and methods Intervention: Participants in the intervention group download a patient supporting app (MyPso SmarTop™ Version 1.0, owned by Leo Pharma) which combined with an EM (SmarTop™ number 053776, owned by Leo Pharma) has three functions: 1) Measures use of medication through EM, 2) measures degree of psoriasis by patients tracking symptoms, and 3) supports the patient with treatment and refill reminders.

Study type: Single-blind block randomized controlled trial. Sampling: Patients are sampled from the dermatology out-patient clinic at Odense University Hospital.

Eligibility criteria: Psoriasis patients aged 18-75 years with mild-moderate psoriasis. It is mandatory that patients have a smartphone and basic skills for use of the smartphone.

Estimated sample size: To be able to improve medical adherence, the investigators wish to detect an 8 % difference between number of applications between intervention and control arm in use of Enstilar© over a 4 week treatment period. Confidence Interval (two-sided) using 95 % C.I., power 80, ratio of sample size 1, mean number of application in intervention Group 90 % of recommended daily application / 4 weeks, S.D. 15 %, drop-outs maximum 10 %:

Total sample size: 134 participants All participants will be seen by trial principal investigator at all of the study visits.

Disclosure and informed signed consent will be obtained before inclusion: The patients are aware they test new equipments, but not informed that they are being monitored or the purpose of the study.

Randomization: Single-blind block randomized controlled trial. Procedure: At the first study visit the trial investigator obtains information regarding gender, age and estimates use of Enstilar© for 4 weeks based on involved Body Surface Area (BSA).

For randomization the investigators use blocks based on 1) age and 2) gender.

Procedures at baseline study visit: While the patient fills the Dermatology Life Quality Index (DLQI) questionnaire, the trial investigator inserts baseline data into the programme REsearch Data Capture (REDCap©) randomize, which randomizes into an intervention- and control arm. Both intervention- and control group receive Enstilar© in the consultation.

To avoid attrition bias from the prescribing doctor, knowledge regarding which patients that are randomized for the intervention is restricted to one nurse until last study visit. After the consultation the patient is referred to a nearby room, where the nurse has access to see into which group the participant has been randomized. If the participant is randomized to the app group, the nurse will instruct the patient in how to download the app on their smartphone and give standard of care instructions regarding how to adhere to the treatment plan. The participants in the control group will reveive standard of care instructions from the nurse regarding how to adhere to the treatment plan. The nurse will not disclose that the patient is being monitored. At the baseline visit the nurse delivers free study medication (Enstilar©) to all participants.

Baseline: Medical history, socio-economic data, DLQI (Dermatology Life Quality Index) and LS-PGA (Lattice System Physician's Global Assessment).

Primary outcome measure week 4: Rate of secondary nonadherence to Enstilar© is obtained using three different Measurements:

Estimated use 0.5 g Enstilar© / % Body Surface Area (BSA) involved / use of Enstilar© in a 4-week treatment period (measured by weight of Enstilar© cans)

Number of estimated applications in the treatment period / Number of Applied applications in the treatment period (measured by EM)

Reported by the patient on an interval scale

Secondary outcome measures week 4, 8, and 26: DLQI and LS-PGA. At study visit week 4 the patients return the EM to the investigator.

Conclusion: If the app for smartphones with the EM can improve adherence and significantly improve secondary outcome measures long-term (week 26), there are promising potentials for implementing the app in the clinic. To the investigators knowledge, this is the first study in topically treated psoriasis, testing if an intervention delivered by in app for smartphones can improve medical adherence.

ELIGIBILITY:
Inclusion Criteria:

* Psoriasis patients aged 18-75 years with mild-moderate psoriasis. It is mandatory that patients have a smartphone and basic skills for use of the smartphone.

Exclusion Criteria:

* aged under 18 and above 75 years, guttate psoriasis, severe degree of psoriasis, i.e. pustular and erythrodermic psoriasis, lack of smartphone and user skills for the smartphone

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2017-01-09 (Actual); Primary Completion 2017-04-29 (Actual); Study Completion 2017-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mathias Tiedemann Svendsen, MD, PhD, Principal Investigator — Department of Dermatology and Allergy Centre, Odense University Hospital
Locations (1):
- Department of Dermatology and Allergy Centre, Odense C, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Svendsen MT, Andersen F, Andersen KH, Andersen KE. Can an app supporting psoriasis patients improve adherence to topical treatment? A single-blind randomized controlled trial. BMC Dermatol. 2018 Feb 7;18(1):2. doi: 10.1186/s12895-018-0071-3. PMID 29415699
- [Result] Svendsen MT, Andersen F, Andersen KH, Pottegard A, Johannessen H, Moller S, August B, Feldman SR, Andersen KE. A smartphone application supporting patients with psoriasis improves adherence to topical treatment: a randomized controlled trial. Br J Dermatol. 2018 Nov;179(5):1062-1071. doi: 10.1111/bjd.16667. Epub 2018 Jul 5. PMID 29654699

RESULTS

PARTICIPANT FLOW:
Groups:
- App as Intervention + Enstilar©: Patients prescribed Enstilar© receive the intervention EM with app for smartphone and conventional instruction from a nurse in the consultation.
  Enstilar 0.005%-0.064% Topical Foam
- Conventional Instructions + Enstilar©: Patients receive conventional instructions from a nurse in the consultation in how to use prescribed Enstilar© with EM.
  Enstilar 0.005%-0.064% Topical Foam
Period: Overall Study
Arm/Group | App as Intervention + Enstilar© | Conventional Instructions + Enstilar©
Started | 68 | 66
Completed | 61 | 61
Not Completed | 7 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | App as Intervention + Enstilar© | Conventional Instructions + Enstilar© | Total
Number analyzed (Participants) | 68 | 66 | 134
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 53 | 53 | 106
  >=65 years | 15 | 13 | 28
Age, Continuous [Mean (Full Range); unit: years] | 50 [23 to 75] | 48 [21 to 72] | 48 [21 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 25 | 52
  Male | 41 | 41 | 82
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Denmark | 68 | 66 | 134

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Adherent Participants
Description: Rate of adherent patients, defined as dichotomized adherence rates obtained by number of days with applied medication with a selected cut-off of 80%, with adherence rates above 80% considered adherent
Time Frame: Week 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | App as Intervention + Enstilar© | Conventional Instructions + Enstilar©
Number analyzed (Participants) | 68 | 66
percentage of participants | 65 [53 to 77] | 38 [26 to 51]
Statistical Analysis 1: Comparison: App as Intervention + Enstilar© vs Conventional Instructions + Enstilar©; Test type: Superiority; p = 0.004, Regression, Logistic; Odds Ratio (OR) = 2.99, 95% CI 2-sided [1.42 to 6.28]

2. Secondary Outcome: Dermatology Life Quality Index (DLQI)
Description: Change from baseline to week 4
  Description of Dermatology Life Quality Index (DLQI): A score from 0-30 [0, patients' quality of life not affected; 30, patients' quality of life severely affected by the skin disease]. The DLQI-scale is a summary of 10 questions on subscales, where patients' report how severely their quality of life has been affected for the last week (patient reported outcome measurements (PROM), each subscale have a score from 0 (not affected by skin disease) to 3 (severely affected by skin disease).
  The minimum score is 0 and the highest score is 30, a high score means worse outcome.
Time Frame: Baseline, week 4, 8 and 26
Population: Patients lost to follow-up
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Conventional Instructions + Enstilar©: Conventional Instructions + Enstilar© Changing from baseline to week 4
- App as Intervention + Enstilar©: App as intervention + Enstilar© Changing from baseline to week 4
Arm/Group | Conventional Instructions + Enstilar© | App as Intervention + Enstilar©
Number analyzed (Participants) | 66 | 68
units on a scale
  Change from baseline to week 4 | 4.54 [3.47 to 5.61] | 4.12 [3.27 to 4.98]
  Change from baseline to week 8: number analyzed (Participants) | 63 | 64
  Change from baseline to week 8 | 5.17 [3.92 to 6.43] | 4.59 [3.71 to 5.48]
  Change from baseline to week 26: number analyzed (Participants) | 61 | 61
  Change from baseline to week 26 | 5.00 [3.69 to 6.31] | 4.23 [3.25 to 5.21]
Statistical Analysis 1: Comparison: Conventional Instructions + Enstilar© vs App as Intervention + Enstilar©; DLQI: Change baseline to week 4; Test type: Superiority; p = 0.545, Regression, Linear; Coefficient = -0.415, 95% CI 2-sided [-1.770 to 0.939]
Statistical Analysis 2: Comparison: Conventional Instructions + Enstilar© vs App as Intervention + Enstilar©; DLQI: Change from baseline to week 4; Test type: Superiority; p = 0.545, Regression, Linear; Coefficient = -0.415, 95% CI 2-sided [-1.770 to 0.939]
Statistical Analysis 3: Comparison: Conventional Instructions + Enstilar© vs App as Intervention + Enstilar©; DLQI: Change from baseline to week 8; Test type: Superiority; p = 0.450, Regression, Linear; Coefficient = -0.581, 95% CI 2-sided [-2.099 to 0.938]
Statistical Analysis 4: Comparison: Conventional Instructions + Enstilar© vs App as Intervention + Enstilar©; DLQI: Change from baseline to week 26; Test type: Superiority; p = 0.348, Regression, Linear; Coefficient = -0.770, 95% CI 2-sided [-2.389 to 0.848]

3. Secondary Outcome: Lattice-System Physician's Global Assessment (LS-PGA)
Description: Change from baseline to week 4, 8 and 26
  Lattice System Physican's Gloabal Assessment (LS-PGA) is a measure from 0-8 (0, patients skin clear; 8, patients' skin severely affected by psoriasis). The scale is a summary of three subscales: 1). thickness of psoriasis, 2). extent of scaling and 3). body surface ares (BSA) affected. The minimum score is 0 and the maximum score is 8, a high score represents a worse outcome.
Time Frame: Week 4, 8 and 26
Population: Lost to follow-up
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Conventional Instructions + Enstilar©: Conventional Instructions + Enstilar© arm changing in LS-PGA form baseline to week 26.
- App + Enstilar©: App + Enstilar© arm changing in LS-PGA from baseline to week 26
Arm/Group | Conventional Instructions + Enstilar© | App + Enstilar©
Number analyzed (Participants) | 66 | 68
units on a scale
  Change from baseline to week 4: number analyzed (Participants) | 65 | 65
  Change from baseline to week 4 | 1.46 [1.17 to 1.75] | 1.86 [1.59 to 2.13]
  Change from baseline to week 8: number analyzed (Participants) | 63 | 64
  Change from baseline to week 8 | 2.16 [1.86 to 2.46] | 2.25 [1.96 to 2.54]
  Change from baseline to week 26: number analyzed (Participants) | 61 | 61
  Change from baseline to week 26 | 1.80 [1.49 to 2.11] | 1.98 [1.66 to 2.31]
Statistical Analysis 1: Comparison: Conventional Instructions + Enstilar© vs App + Enstilar©; LS-PGA: Change from baseline to week 4; Test type: Superiority; p = 0.047, Regression, Linear; coefficient = 0.400, 95% CI 2-sided [0.005 to 0.795]
Statistical Analysis 2: Comparison: Conventional Instructions + Enstilar© vs App + Enstilar©; LS-PGA: Change from baseline to week 8; Test type: Superiority; p = 0.662, Regression, Linear; Coefficient = 0.091, 95% CI 2-sided [-0.321 to 0.504]
Statistical Analysis 3: Comparison: Conventional Instructions + Enstilar© vs App + Enstilar©; LS-PGA: Change from baseline to week 26; Test type: Superiority; p = 0.424, Regression, Linear; Coefficient = 0.180, 95% CI 2-sided [-0.264 to 0.625]

ADVERSE EVENTS:
Time Frame: Information on adverse events systematically reported at visits at baseline, week 4, 8 and 26 (6 months)
Groups:
- Conventional Instructions + App as Intervention + Enstilar©; App as Intervention + Enstilar©: Information obtained baseline, week 4, 8 and 26.
  Participants were treated with Enstilar© once daily when needed for 6 months
Arm/Group | Conventional Instructions + App as Intervention + Enstilar© | App as Intervention + Enstilar©
All-Cause Mortality (participants affected / at risk) | 0/66 | 0/68
Serious Adverse Events (participants affected / at risk) | 0/66 | 1/68
Other Adverse Events (participants affected / at risk) | 22/66 | 20/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Conventional Instructions + App as Intervention + Enstilar© (N=66) | App as Intervention + Enstilar© (N=68)
Infection in knee prosthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Infection in knee prosthesis. Not Associated with the use of Cal/BD foam.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Conventional Instructions + App as Intervention + Enstilar© (N=66) | App as Intervention + Enstilar© (N=68)
relapse of carcinoma in situ of the glottis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) — Not related to use of Cal/BD foam
Worsening of chronic obstructive pumonary disease (COPD) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Associated to accidentally inhaling gas from canister containing Cal/BD foam
Nausea (Ear and labyrinth disorders) | 2 (2) | 1 (1)
Elevated liver enzymes (Hepatobiliary disorders) | 2 (2) | 1 (1) — Elevated liver enzymes after treatment with methotrexate. Not related to use of Cal/BD foam
Elevated creatinin levels (Renal and urinary disorders) | 0 (0) | 1 (1)
Skin manifestations (Skin and subcutaneous tissue disorders) | 8 (8) | 8 (8) — 11 different skin manifestations not directly related to use of Enstilar
various musculoskelatal disorders (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (4) — Not related to the use of Cal/BD foam
Fainting (Vascular disorders) | 1 (1) | 0 (0) — Fainting not related to use of Cal/BD foam
Lung and skin infections (Infections and infestations) | 4 (4) | 4 (4) — Not related to the use of Cal/BD foam

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-03): https://cdn.clinicaltrials.gov/large-docs/13/NCT02858713/Prot_SAP_000.pdf